CLINICAL TRIAL: NCT05302193
Title: Non-invasive Blood Pressure Measurement Using Samsung Smartwatch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NIBPsmartwatch21
Record Dates: First submitted 2022-03-16; First posted 2022-03-31 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Blood Pressure; Heart Rate
Keywords: blood pressure measurement; heart rate measurement; smartwatch
MeSH Terms: interventions — Heart Rate; Exercise

STUDY DESIGN:
Intervention Model Description: Two measuring devices are active simultaneously during measurement of blood pressure and heart rate on each participant and their functioning is compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood pressure and heart rate measurement (Experimental): Calm measurement of blood pressure and heart rate simultaneously by smartwatch and vital signs monitor. Each participant will undergo this measurement a total of 6 times.
  Interventions: Other: Calm measurement of blood pressure and heart rate (before physical activity); Other: Physical activity; Other: Calm measurement of blood pressure and heart rate (after physical activity)

INTERVENTIONS:
Other: Calm measurement of blood pressure and heart rate (before physical activity) — Simultaneous blood pressure and heart rate measurements at minutes 2 and 5.5 of the experiment.
Other: Physical activity — Five minutes of physical activity, between times 7.5 min and 12.5 min of the experimental part. Riding on a spinning ergometer with a standardized load of 1 W/kg.
Other: Calm measurement of blood pressure and heart rate (after physical activity) — Simultaneous blood pressure and heart rate measurements at times 15.5, 17, 20.5 and 22 minutes of the experimental part.

SUMMARY:
The aim of this study is to verify the accuracy of blood pressure and heart rate measurement by Samsung smartwatches compared to a standard monitor of vital signs used in intensive care units.

DETAILED DESCRIPTION:
Recently, wearables, like smartwatches, have been gaining new possibilities in monitoring biological signals and they are used for home monitoring of health conditions. Heart rate measurement is a common function of smartwatches, some smartwatch models even measure blood pressure. The study aims to compare the measurement of blood pressure and heart rate using the latest smartwatch with a vital signs monitor used in clinical practice. Blood pressure and heart rate measurements will be taken by hand from the watch and the vital signs monitor simultaneously. The agreement of the measurements of both devices will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* any acute illness
* pregnancy
* severe cardiovascular conditions
* severe asthma or other severe respiratory conditions
* diabetes
* hypotension or hypertension

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Similarity of blood pressure measurements from two devices | 1 hour
  The agreement of systolic and diastolic blood pressure measurements of both monitoring devices will be evaluated.
Similarity of heart rate measurements from two devices | 1 hour
  The agreement of heart rate measurements of both monitoring devices will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Rafl Huttova, MSc, Principal Investigator — Czech Technical University in Prague; Jakub Rafl, PhD, Principal Investigator — Czech Technical University in Prague; Martin Rozanek, PhD, Principal Investigator — Czech Technical University in Prague
Locations (1):
- Faculty of Biomedical Engineering, Czech Technical University in Prague, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hahnen C, Freeman CG, Haldar N, Hamati JN, Bard DM, Murali V, Merli GJ, Joseph JI, van Helmond N. Accuracy of Vital Signs Measurements by a Smartwatch and a Portable Health Device: Validation Study. JMIR Mhealth Uhealth. 2020 Feb 12;8(2):e16811. doi: 10.2196/16811. PMID 32049066